CLINICAL TRIAL: NCT06335836
Title: The Effects of Social Isolation and Social Interaction on the Risk of Dementia Progression and Brain Function in SCD (Subjective Cognitive Decline, SCD)
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-127; 2024-SR-127 (Other: Ethics Committee of Nanjing Medical University)
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Social Isolation; SCD; Subjective Cognitive Decline; MCI; Mild Cognitive Impairment; AD; Alzheimer Disease
MeSH Terms: conditions — Social Isolation; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — venous blood： amyloid tau APOE genotyping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SI group (social isolation group): The LSNS-6 was used for assessing social networks among older Chinese. Lubben suggested using a score of less than 12 as a clinical cutoff point of the LSNS-6 to indicate social isolation, which meant, on average, the respondents had less than two people to perform social integration functions.
  0≤LSNS-6≤12
  Interventions: Behavioral: social isolation
- nonSI group (non-social isolation group): LSNS-6>12

INTERVENTIONS:
Behavioral: social isolation — social isolation (0≤LSNS-6≤12)
  Groups: SI group (social isolation group)

SUMMARY:
The goal of this clinical trial is to learn about the effects of social isolation and social interaction on the risk of dementia progression and brain function in SCD

1. To explore the association between social isolation and lonely SCD populations and the occurrence and progression of MCI and AD through cross-sectional studies, cohort studies and randomized controlled trials of SCD;
2. To clarify the correlation between different carrier states, resting brain function connectivity characteristics, and dual-task walking ability of APOEε4 allele and the progression of SCD to MCI and AD during the cognitive progress of people with SCD affected by social isolation;
3. Establish a predictive model of cognitive decline from SCD to MCI and AD, and apply it to the SCD population to carry out individualized interventions;
4. Confirm the protective effect of social interaction on cognitive level and brain function in SCD patients.

DETAILED DESCRIPTION:
1. to explore the impact of social isolation on the risk of progression to MCI or AD in the SCD population.

1. A cohort study design was enrolled in the SCD population, assess the degree of social isolation, and analyze the impact of social isolation, an exposure factor, on the progression of SCD patients to MCI or AD by collecting 3-5 years follow-up data;
2. To analyze the interaction between the degree of social isolation of SCD patients and the connectivity characteristics of executive control, default network, and language network in the brain functional network.

2. the predictive effects of APOE-ε4 genotype, degree of social isolation, loneliness, and dual-task walking ability on the risk of SCD progression to MCI and AD in SCD population.

1. Using data from a cohort study, a prediction model of the SCD population with APOE-ε4 genotype, degree of social isolation, loneliness, dual-task walking parameter, degree of executive-control brain network connectivity, and degree of depression was developed to predict the risk of SCD progression to MCI and AD;
2. Use the above prediction model to apply to the clinic for prognostic prediction and individualized risk factor control in the SCD population.

ELIGIBILITY:
Inclusion Criteria:

* SCD

  1. Self-perceived continuous cognitive decline compared with the previous normal state, and is not related to acute events;
  2. After adjustment for age, gender, and years of education, the standard cognitive test is normal, or the diagnostic criteria for MCI are not met;
  3. Selected candidates can sign the informed consent form themselves.

Exclusion Criteria:

* (a) Aged under 45 years or older than 85 years; (b) Vascular dementia or other central nervous system diseases; (c) Hachinski Ischemic Scale score > 4 points; (d); Unable to complete neuropsychological tests (e.g., blindness, deafness, severe language impairment); (e) Drug abuse or alcohol dependency within the last 6 months; (f) Current participation in other cognition studies; (g) Severe diabetes mellitus, or severe cardiovascular disease, cerebrovascular disease, liver diseases, kidney diseases, psychiatric disorders; (h) Contraindications to imaging techniques: claustrophobia, metallic implants (e.g., intracranial metal clips), electronic devices (e.g., cardiac pacemakers)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were grouped as SCD when they reported cognitive decline compared with a previous state, whereas neuropsychological battery and other objective investigations (adjusted age, gender, and education) were normal, and criteria for MCI, dementia, or any other neurologic or psychiatric diseases that potentially cause cognitive complaints were not met.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Mild Cognitive Impairment (MCI) | through study completion, an average of 1 year
  Incidence of Mild Cognitive Impairment (MCI)
Incidence of Alzheimer's disease (AD) | through study completion, an average of 1 year
  Incidence of Alzheimer's disease (AD)

SECONDARY OUTCOMES:
AVLT-H | through study completion, an average of 1 year
  Auditory Verbal Learning Test Huashan Version, AVLT-H The Auditory Verbal Learning Test-Huashan version (AVLT-H) assessment will be used as the primary outcome to assess EM for our study. The AVLT-H assesses several aspects of verbal EM through a list of 12 words, such as short or long-term delayed recall and recognition. It has been widely used as a semantic categorization memory test in mainland Chinese populations.
MoCA | through study completion, an average of 1 year
  Montreal Cognitive Assessment, MoCA Overall cognitive function will be assessed using scores from the Montreal Cognitive Assessment Test (MOCA).
WMS-RLM | through study completion, an average of 1 year
  Wechsler Memory Scale-Revised Logical Memory, WMS-RLM Participants were asked to recall the stories they had heard after listening to a short story containing 25 information points, with 1 point for each information point and 25 points for each story, for a total of two stories out of 50 points, with higher scores indicating better short-term memory.
WDS | through study completion, an average of 1 year
  Wechsler Digit Span, WDS The scale is divided into two parts, forward numerical memory and inverse numerical memory, with 12 items each, with a maximum of 12 points and a maximum score of 24 points, with higher scores leading to better short-term memory and attention.
VFT | through study completion, an average of 1 year
  Verbal Fluency Test, VFT This scale is a measure of verbal fluency and requires the test subject to say as many names as possible in one minute, with only one repeat counted and the total number recorded.
BNT | through study completion, an average of 1 year
  Boston Naming Test, BNT This scale, one of the most commonly used methods for diagnosing naming disorder, consists of 30 black-and-white pictures of objects commonly used in daily life, and the test subjects are asked to name the pictures and record the total number of correct responses.
LSNS-6 | through study completion, an average of 1 year
  Lubben Social Network Scale-6, LSNS-6 The LSNS-6 could be a useful tool for assessing social networks among older mainland Chinese. In addition, suggestion is made to improve social networks, especially in family bonds and support, as a promising strategy in reducing late-life suicide risks in mainland China.
UCLA | through study completion, an average of 1 year
  UCLA Loneliness Scale, University of California at Los Angels The 20-item UCLA Loneliness Scale (Version 3; UCLA-3) is a commonly used assessment of loneliness, with strong test-retest reliability as well as high internal consistency and validity (Cronbach's α of .89 to .94).
GDS | through study completion, an average of 1 year
  Geriatric Depression Scale, GDS Participants completed the short form of the Geriatric Depression Scale (GDS), a 15-item assessment to screen for depression in older adults, with higher scores indicating greater severity.
PSQI | through study completion, an average of 1 year
  Pittsburgh sleep quality index, PSQI Self-reported sleep quality was assessed using the Pittsburgh Sleepiness Quality Index (PSQI).
DTC | through study completion, an average of 1 year
  Dual task consumption, DTC Dual-task cost (DTC) is the percentage change in walking speed between single-task and dual-task. It has been suggested that DTC predicts the risk of progression to dementia in older patients with MCI, with higher DTC and shorter time to progression to dementia and a higher risk.
fMRI | Enrollment, 3, 5 years later
  fMRI
tau | Enrollment, 3, 5 years later
  tau
Aβ | Enrollment, 3, 5 years later
  Aβ
APOE genotyping | Enrollment
  APOE genotyping Genotypes for rs7412 and rs429358, the single nucleotide polymorphisms (SNPs) defining the ϵ-2, ϵ-3 and ϵ-4 alleles of APOE, were genotyped using the commercially available TaqMan® SNP Genotyping Assay (ThermoFisher Scientific).
TMT-A, TMT-B | through study completion, an average of 1 year
  The online test is a connected test (Chinese revised version), and the test is divided into two parts, A and B, each of which includes exercises and tests. Before taking the test, the test taker should be asked to practice and then take the assessment. TMT-A requires the test subject to complete the connection from 1 to 25 as quickly as possible, in the order from smallest to largest, and the pen must not leave the paper during the connection. TMT-B requires the test subject to complete the connection from 1 to 25 as quickly as possible in the order of small to large, circle icon and square icon interval, and the pen must not leave the paper during the connection process. The time spent in each of the two parts is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Yi, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China, Jiangsu, China